CLINICAL TRIAL: NCT03453359
Title: Bispectral Index Monitoring for Sedation in Elective Colonoscopies of Adult Patients: a Randomized Controlled Trial
Acronym: BIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Galdakao-Usansolo (Other Government)
Responsible Party: Principal Investigator, Iratxe González Mendibil, Principal Investigator, Hospital Galdakao-Usansolo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 01/18
Record Dates: First submitted 2018-01-27; First posted 2018-03-05 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Colonoscopy
Keywords: bispectral index monitor; sedation; adverse effects

STUDY DESIGN:
Intervention Model Description: We compared the results of two groups of patients. Experimental group, in which sedation is adjusted using as main parameters the information obtained by the bispectral index monitor. Control Group, with sedation based on subjective monitoring using the Ramsay scale as a reference.
Who Masked: Participant, Care Provider
Masking Description: Patients will be randomly assigned to one of the two study groups. The anesthesiologist who records the information knows which group they belong to, according to a randomization table provided in collaboration with the Research Unit, but the patients do not know it.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BIS (Experimental): Group of patients (90) in whom sedation is adjusted using as main parameters the information obtained by the BIS sedation monitor (BIS VISTA, Aspect Medical Systems, USA).
  Interventions: Device: BIS monitor
- Ramsay (Active Comparator): Group of patients (90) in whom sedation is based on subjective monitoring of the level of sedation, using the Ramsay scale as a reference.
  Interventions: Device: Ramsay scale

INTERVENTIONS:
Device: BIS monitor — The investigators will place on the forehead of all patients the sensor BIS quatroTM, that connects with this monitor, and they will guide sedation and will record the values obtained.
  Other Names: BIS VISTA; Aspect Medical Systems, USA
  Arms: BIS
Device: Ramsay scale — In this group, sedation is guided by the Ramsay monitoring scale. The investigators will talk with the patients and will determine the corresponding level of sedation.
  Other Names: Conventional monitoring
  Arms: Ramsay

SUMMARY:
The primary aim of the study is to determine the rate sedation-induced adverse events, comparing BIS-guided sedation with clinical observation. Secondary outcomes were to examine patient characteristics who developed adverse events, propofol and remifentanil dosage and patient satisfaction analyzing different time points undergoing elective colonoscopy.

DETAILED DESCRIPTION:
Randomized double-blind clinical trial in patients undergoing scheduled colonoscopies in endoscopy rooms of the Galdakao-Usánsolo Hospital (Bizkaia, Spain) and Mendaro Hospital (Gipuzkoa, Spain). The investigators will compare the rate of cardiorrespiratory adverse events as well as the anesthetic drugs dosage, need for rescue medication and patient satisfaction among the experimental group in which sedation is guided by BIS and the control group in which the anesthesiologist is blind to the result of the BIS. The investigators hypothesized that BIS monitoring would be associated with better outcomes than clinical observation.

The BIS is the parameter of anesthetic depth monitoring most used today. Its use was approved by the Food and Drug Administration (FDA) in 1996 as an aid to control the effects of certain anesthetic agents. It is validated in the operating room (Recommendation grade A), but not outside it due to lack of conclusive studies.

180 patients are needed to obtain statistically significant differences between both groups. Qualitative variables are expressed in the form of frequencies and percentages and continuous variables in the form of means and standard deviations. Comparisons of percentages will be made by the Chi square test (or Exact Fisher's test, when the expected frequencies are less than 5) and the difference of means in the continuous variables by the t test as well as by the Wilcoxon nonparametric test if the distribution of the variable requires it. The degree of agreement between the BIS and Ramsay scale will be made through the weighted Kappa test. Statistical significance will be assumed when p <0.05. All statistical analyzes will be carried out using SAS V9.4. (SAS institute, Inc., Carey, NC).

ELIGIBILITY:
Inclusion Criteria:

* Indication of complete colonoscopy on a scheduled basis.
* Classification of physical status ASA I, II and III, with the exception of patients with moderate to severe kidney and / or liver disease.
* Intermittent or persistent mild asthma. It implies the absence of daily symptoms and FEV1> 80% (GINA 2004).
* Body Mass Index (BMI) less than 35 kg / m2, and greater than 18 kg/m2.
* Intact neurological capacity.
* Acceptance to participate in the study after the contribution of written informed consent.

Exclusion Criteria:

* ASA IV.
* BMI greater than 35 kg / m2, and less than 18 kg/m2.
* Refusal to participate in the study.
* Allergy to any of the medications used in sedation, or its components.
* Known mental or neurological disease.
* Renal and / or moderate to severe Hepatic insufficiency.
* Chronic Obstructive Pulmonary Disease (COPD) or Obstructive Sleep Apnea.
* Chronic opiate users.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2018-01-28 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Sedation-induced adverse events | 1 year.
  Compare the rate of cardiorrespiratory adverse events between the two groups

SECONDARY OUTCOMES:
Characteristics of patients who developed adverse events | 1 year.
  Describe the patient characteristics
The pharmacological dosage | 1 year.
  The investigators will note if there is significant differences in the dose of phamacological drugs, and rescue propofol
Level of satisfaction with the colonoscopy. | 1 year.
  The investigators will distribute a satisfaction questionnaire to all patients after the colonoscopy to find out their opinion about the quality of sedation.

CONTACTS AND LOCATIONS:
Overall Officials: Iratxe Gonzalez Mendibil, MD, Principal Investigator — Hospital Galdakao-Usansolo
Locations (1):
- Hospital Galdakao-Usansolo, Galdakao, Vizcaya, Spain

IPD SHARING:
Plan to Share IPD: Yes
The investigators have a randomization table to assign the intervention of each patient. The investigators will record anthropometric data and the parameters resulting from the monitoring. These data will be available to collaborating investigators and subsequently to a member of the Research Unit who will record this information in a database that will be analyzed to obtain results.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: This study will begin in January 2018 and will end after the recruitment of the 180 patients and subsequent data analysis, approximately in June 2020.
Access Criteria: The Principal Investigator has produced an Information Manual for collaborators where the protocol and the objectives of the study are detailed. This information has been sent via email and is printed and available in the endoscopy room where the registration will take place. The information folder includes the randomization table, informed consent, patient information sheet, data record sheet and record sheet for the BIS parameters of the patients in the Ramsay group. This information has been transmitted orally and an informative session has been held for all the members of the project.
  Members of the Research Unit will perform a check of this information, correlating it with what is described in the anesthesia chart and reviewing the patient data in the health system database. In addition, they will collaborate with the statistical analysis and obtaining results.

REFERENCES:
- [Background] Thomson A, Andrew G, Jones DB. Optimal sedation for gastrointestinal endoscopy: review and recommendations. J Gastroenterol Hepatol. 2010 Mar;25(3):469-78. doi: 10.1111/j.1440-1746.2009.06174.x. PMID 20370725
- [Background] Dumonceau JM, Riphaus A, Schreiber F, Vilmann P, Beilenhoff U, Aparicio JR, Vargo JJ, Manolaraki M, Wientjes C, Racz I, Hassan C, Paspatis G. Non-anesthesiologist administration of propofol for gastrointestinal endoscopy: European Society of Gastrointestinal Endoscopy, European Society of Gastroenterology and Endoscopy Nurses and Associates Guideline--Updated June 2015. Endoscopy. 2015 Dec;47(12):1175-89. doi: 10.1055/s-0034-1393414. Epub 2015 Nov 12. No abstract available. PMID 26561915
- [Background] Park WY, Shin YS, Lee SK, Kim SY, Lee TK, Choi YS. Bispectral index monitoring during anesthesiologist-directed propofol and remifentanil sedation for endoscopic submucosal dissection: a prospective randomized controlled trial. Yonsei Med J. 2014 Sep;55(5):1421-9. doi: 10.3349/ymj.2014.55.5.1421. PMID 25048506
- [Background] Hong MJ, Sung IK, Lee SP, Cheon BK, Kang H, Kim TY. Randomized comparison of recovery time after use of remifentanil alone versus midazolam and meperidine for colonoscopy anesthesia. Dig Endosc. 2015 Jan;27(1):113-20. doi: 10.1111/den.12383. Epub 2014 Nov 11. PMID 25251893
- [Background] Lera dos Santos ME, Maluf-Filho F, Chaves DM, Matuguma SE, Ide E, Luz Gde O, de Souza TF, Pessorrusso FC, de Moura EG, Sakai P. Deep sedation during gastrointestinal endoscopy: propofol-fentanyl and midazolam-fentanyl regimens. World J Gastroenterol. 2013 Jun 14;19(22):3439-46. doi: 10.3748/wjg.v19.i22.3439. PMID 23801836
- [Background] Yu YH, Han DS, Kim HS, Kim EK, Eun CS, Yoo KS, Shin WJ, Ryu S. Efficacy of bispectral index monitoring during balanced propofol sedation for colonoscopy: a prospective, randomized controlled trial. Dig Dis Sci. 2013 Dec;58(12):3576-83. doi: 10.1007/s10620-013-2833-4. Epub 2013 Aug 28. PMID 23982208
- [Background] Sasaki T, Tanabe S, Azuma M, Sato A, Naruke A, Ishido K, Katada C, Higuchi K, Koizumi W. Propofol sedation with bispectral index monitoring is useful for endoscopic submucosal dissection: a randomized prospective phase II clinical trial. Endoscopy. 2012 Jun;44(6):584-9. doi: 10.1055/s-0032-1306776. Epub 2012 May 25. PMID 22638779
- [Background] Imagawa A, Fujiki S, Kawahara Y, Matsushita H, Ota S, Tomoda T, Morito Y, Sakakihara I, Fujimoto T, Taira A, Tsugeno H, Kawano S, Yagi S, Takenaka R. Satisfaction with bispectral index monitoring of propofol-mediated sedation during endoscopic submucosal dissection: a prospective, randomized study. Endoscopy. 2008 Nov;40(11):905-9. doi: 10.1055/s-2008-1077641. PMID 19023932
- [Background] Qadeer MA, Vargo JJ, Patel S, Dumot JA, Lopez AR, Trolli PA, Conwell DL, Stevens T, Zuccaro G Jr. Bispectral index monitoring of conscious sedation with the combination of meperidine and midazolam during endoscopy. Clin Gastroenterol Hepatol. 2008 Jan;6(1):102-8. doi: 10.1016/j.cgh.2007.10.005. Epub 2007 Dec 11. PMID 18065278
- [Background] Liu SS. Effects of Bispectral Index monitoring on ambulatory anesthesia: a meta-analysis of randomized controlled trials and a cost analysis. Anesthesiology. 2004 Aug;101(2):311-5. doi: 10.1097/00000542-200408000-00010. PMID 15277912
- [Background] Bower AL, Ripepi A, Dilger J, Boparai N, Brody FJ, Ponsky JL. Bispectral index monitoring of sedation during endoscopy. Gastrointest Endosc. 2000 Aug;52(2):192-6. doi: 10.1067/mge.2000.107284. PMID 10922090
- [Background] Oliveira CR, Bernardo WM, Nunes VM. Benefit of general anesthesia monitored by bispectral index compared with monitoring guided only by clinical parameters. Systematic review and meta-analysis. Braz J Anesthesiol. 2017 Jan-Feb;67(1):72-84. doi: 10.1016/j.bjane.2015.09.001. Epub 2016 Apr 14. PMID 28017174

DOCUMENTS (2):
  • Study Protocol (2018-01-28): https://cdn.clinicaltrials.gov/large-docs/59/NCT03453359/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-28): https://cdn.clinicaltrials.gov/large-docs/59/NCT03453359/SAP_001.pdf